CLINICAL TRIAL: NCT06121726
Title: Evaluation of Predictive Factors for the Effectiveness of the Ilioinguinal Iliohypogastric Nerve Block in Unilateral Inguinal Hernioplasty
Brief Title: Predictive Factors for the Effectiveness of the Ilioinguinal Iliohypogastric Nerve Block for Hernia Surgery
Acronym: VALI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, MD, University of Padova
Other Study IDs: VALI
Record Dates: First submitted 2023-10-13; First posted 2023-11-08 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Hernia Inguinal; Pain Postoperative; Regional Anesthesia
Keywords: ilioinguinal; iliohypogastric; nerve block; pain; hernia
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Pain; Hernia | interventions — Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ilioinguinal-Iliohypogastric nerve block: Patients will receive Ilioinguinal-Iliohypogastric nerve block as standard of care
  Interventions: Other: Ilioinguinal-Iliohypogastric nerve block; Drug: Local anesthetic

INTERVENTIONS:
Other: Ilioinguinal-Iliohypogastric nerve block — local anesthetic will be administered near ilioinguinal-iliohypogastric nerves under ultrasound guidance. Given the observational nature of the study dose and drugs will be decided by the attending anesthesiologist
Drug: Local anesthetic — Given the observational nature of the study dose and drugs will be decided by the attending anesthesiologist

SUMMARY:
Inguinal hernia repair is a common surgical procedure done as day surgery. Because patients need to be discharged on the same day, the choice of anesthesia technique is influenced. One option is the ilioinguinal (II)-iliohypogastric (IH) nerve block, a type of transversus abdominis plane (TAP) block, which has benefits such as faster recovery, better pain control, and reduced opioid use. It also allows for quick discharge, early feeding, and no need for post-anesthesia or recovery unit stay.

This study aims to evaluate the success of the II-IH nerve block as the preferred anesthesia strategy for patients undergoing unilateral inguinal hernia repair using the Lichtenstein technique. The study will analyze various factors such as BMI, age, optimal ultrasound vision, amount of anesthesia used, dose of anesthesia administered, time between block execution and incision, and sedative dose needed to determine independent variables of block effectiveness.

The study will include patients aged 18 or older, with ASA I-II-III classification, and who provide informed consent. Patients with allergies to local anesthetics, certain medical conditions, obesity, difficulty visualizing target structures, non-cooperative behavior, or taking anticoagulant therapy will be excluded.

The study will be conducted at the Sant'Antonio Hospital (Padova University Hospital) operating rooms for one year, aiming to recruit around 400 patients.

Informed consent for data processing will be obtained during the preoperative anesthesia visit, and standard anesthesia procedures will be followed during the surgery.

As usual care the patient will be monitored before surgery using an electrocardiogram, oxygen saturation measurement, and non-invasive blood pressure. After adequate sedation, the II-IH nerve block will be performed under sterile conditions and ultrasound guidance.

Participation in the study does not modify the commonly used anesthesia procedures and does not pose any additional risks or provide direct benefits to the patients. The data collected will be treated confidentially and used exclusively for the study's purposes.

Data collection will be conducted through a paper-based form, and only a few variables will be recorded. The study's findings will be made public, even if negative, and will be submitted to the ethics committee within twelve months of data collection completion.

DETAILED DESCRIPTION:
Inguinal hernioplasty is one of the most commonly performed surgical procedures in day surgery. The need to discharge the surgical patient on the same day affects the choice of anesthetic strategy and leads to opt for those techniques that allow for faster recovery. One option is represented by the ilioinguinal (II)-iliohypogastric (IH) nerve block, a variant of the transversus abdominis plane (TAP) block, which has a safety profile, ease of execution, effectiveness in controlling intra- and post-operative pain, with a reduction in opioid administration and increased patient satisfaction. It also has additional advantages, such as rapid patient discharge, early refeeding, no need for post-anesthesia care unit (PACU) or recovery room admission.

It is not yet established what the success rate of the anesthetic block is, intended as the absence of the need for further infiltration by the surgeon, the administration of opioid drugs, or the need to convert to general anesthesia, nor what the independent risk factors are for the positive outcome of the procedure. The aim of this study is therefore to evaluate the success of the ilioinguinal-iliohypogastric block as the anesthetic strategy of choice in patients undergoing unilateral inguinal hernioplasty with the Lichtenstein technique, and the independent variables of block effectiveness, analyzing various parameters such as BMI, age, optimal ultrasound visualization, volume of anesthetic used, dose of anesthetic administered, time elapsed between the execution of the II-IH block and the incision, and the necessary dose of sedative drugs.

All patients who need to undergo unilateral inguinal hernioplasty according to the Lichtenstein technique, aged ≥ 18 years, American Society of Anesthesiology-Physical Status (ASA-PS) I-II-III, and who give their informed consent to participate in the study will be recruited. Patients with allergies to local anesthetics; heart disease, kidney disease, liver disease, uncompensated central or peripheral neuropathy; history of coagulopathy (risk/benefit ratio to be evaluated); infection at the site of the procedure; obesity (high BMI) or difficulty in visualizing target structures will be excluded. Non-cooperative patients or those taking anticoagulant therapy will also not be included.

This observational, prospective, monocentric study will be conducted in the operating rooms of the Sant'Antonio Hospital (Hospital-University Company of Padova) and will last for one year. An attempt will be made to recruit the largest number of patients within this time frame, and considering the surgical activity at the operating facility, it is estimated that approximately 400 patients will be enrolled.

The patient will be recruited after verifying the inclusion/exclusion criteria. Each patient will be informed about the study and asked for written informed consent for the treatment of personal data at the time of the standard preoperative anesthesiology visit.

The intraoperative management of the patient will be at the discretion of the anesthesiologist in charge of the patient, without making any changes to their conduct.

The patient will be monitored in the preoperative room with electrocardiogram, pulse oximetry, and non-invasive blood pressure. Once the patient is positioned on the operating table, after adequate sedation with Propofol Targeted Controlled Infusion, the locoregional anesthesia, or II-IH nerve block, will be performed using a sterile technique and under ultrasound guidance. At the end of the procedure, Paracetamol 1 g will be administered.

With this study, the commonly used anesthetic procedures are not modified, and therefore participation in this study does not entail any additional risk for the patient and there are no direct benefits associated with it. All the clinical activities foreseen for the study are classified as routine procedures as they would be performed or prescribed to the patient even in the event of refusal to participate in the study.

The project's data collection form (CRF) will be paper-based and few variables are expected to be collected. Following the longitudinal design of the study, the CRF will collect data on patients at the time of the anesthesiology visit, during the execution of the II-IH nerve block, and during the surgical procedure. The collected data will be entered into an Excel file by the experimenter and will be processed for the exclusive purposes related to the completion of this study, made anonymous, and, in this form, aggregated in the project's database, solely for the purpose of carrying out the study itself and achieving the predefined objectives. The data will not be disseminated unless in strictly anonymous and aggregated form.

All statistical analyzes will be performed using R version 3.4.0 (2017-04-21). Results will be considered statistically significant for P values ≤ 0.05.

The study data will be made public even in the case of negative results and will be sent in copy to the ethics committee within twelve months from the conclusion of data collection.

ELIGIBILITY:
Inclusion Criteria

* >18 years old
* Informed consent
* Unilateral inguinal hernioplasty program using the Lichtenstein technique

Exclusion criteria

* Allergy to local anesthesia
* Cardiac, renal, hepatic, central or peripheral neuropathies that are not compensated
* Anticoagulant therapy
* History of coagulopathy (evaluate risk/benefit ratio)
* Infection at the surgical site
* Non-cooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing unilateral inguinal hernioplasty
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Described as the need of additional local anesthetic, additional opioids and/or general anesthesia

SECONDARY OUTCOMES:
Total body weight (kg) as predictive parameter for ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Total body weight (kg) as predictive parameter for ilioinguinal-iliohypogastric nerve block failure
Time From Block To Skin Incision(minutes) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Time From Block To Skin Incision(minutes) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure
Dose of anesthetic(mg) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Dose of anesthetic(mg) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure
Local anesthetic volume(mL) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Local anesthetic volume(mL) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure
Age(years) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Age(years) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure
Ultrasound Nerves Visualization (yes/no) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure | through surgery completation, an average of 1 hour
  Ultrasound Nerves Visualization (yes/no) As Predictive Parameter For ilioinguinal-iliohypogastric nerve block failure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: No